CLINICAL TRIAL: NCT00864682
Title: Propofol Mixed With Lidocaine Versus Lidocaine Pretreatment With Tourniquet for Alleviation of Pain Associated With Propofol Injection
Brief Title: Preventing Propofol-associated Injection Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Benaroya Research Institute (Other)
Responsible Party: Principal Investigator, Joseph Neal, PI, Benaroya Research Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 06091
Record Dates: First submitted 2009-03-16; First posted 2009-03-19 (Estimated); Results first posted 2009-08-03 (Estimated); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Pain
Keywords: propofol; lidocaine; injection pain
MeSH Terms: conditions — Pain | interventions — Sodium Chloride; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): Saline pretreatment, saline admixture
  Interventions: Drug: Saline
- Lidocaine pretreatment (Active Comparator): Lidocaine pretreatment / saline-propofol admixture
  Interventions: Drug: lidocaine pretreatment
- Lidocaine-Propofol admixture (Active Comparator): saline pretreatment / Lidocaine-propofol admixture
  Interventions: Drug: Lidocaine / propofol admixture

INTERVENTIONS:
Drug: Saline — 3.3 mL normal saline
  Arms: Placebo
Drug: Lidocaine / propofol admixture — lidocaine 50 mg plus propofol 50 mg intravenous (iv)
  Arms: Lidocaine-Propofol admixture
Drug: lidocaine pretreatment — lidocaine 50 mg iv under tourniquet-control
  Arms: Lidocaine pretreatment

SUMMARY:
Injection of propofol is associated with discomfort in subsets of patients. Local anesthetics have been shown to attenuate this response in some patients. This randomized, double-blind, placebo-controlled trial tests the hypothesis that lidocaine mixed with propofol will be superior to lidocaine administered directly into the vein, under tourniquet control, prior to injection of propofol. Both groups are expected to be superior to placebo.

ELIGIBILITY:
Inclusion criteria:

* weight >40kg, <100kg
* ambulatory surgery

Exclusion criteria:

* allergy to propofol or lidocaine
* taking opioids, benzodiazepines, or nonsteroidal antiinflammatory drugs (NSAIDs)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2008-01; Primary Completion 2009-03 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph M Neal, MD, Principal Investigator — Virginia Mason Medical Center
Locations (1):
- Benaroya Research Institute, Seattle, Washington, United States

REFERENCES:
- [Derived] Walker BJ, Neal JM, Mulroy MF, Humsi JA, Bittner RC, McDonald SB. Lidocaine pretreatment with tourniquet versus lidocaine-propofol admixture for attenuating propofol injection pain: a randomized controlled trial. Reg Anesth Pain Med. 2011 Jan-Feb;36(1):41-5. doi: 10.1097/AAP.0b013e31820306da. PMID 21455088

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients entered were recruited between January 2008 and March 2009. Hospital / ambulatory surgery setting
Groups:
- Control Arm: saline pretreatment, saline plus propofol admixture
- Lidocaine / Propofol Admixture Arm: saline pretreatment, lidocaine plus propofol admixture
- Lidocaine Pretreatment Arm: lidocaine pretreatment, saline plus propofol admixture
Period: Overall Study
Arm/Group | Control Arm | Lidocaine / Propofol Admixture Arm | Lidocaine Pretreatment Arm
Started | 52 | 51 | 53
Completed | 50 | 50 | 51
Not Completed | 2 | 1 | 2
Not completed — Protocol Violation | 2 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Arm | Lidocaine / Propofol Admixture Arm | Lidocaine Pretreatment Arm | Total
Number analyzed (Participants) | 52 | 51 | 53 | 156
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 42 | 41 | 38 | 121
  >=65 years | 10 | 10 | 15 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 53 (14) | 54 (14) | 52 (17) | 53 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 23 | 26 | 79
  Male | 22 | 28 | 27 | 77
Region of Enrollment [Number; unit: participants]
  United States | 52 | 51 | 53 | 156.0

OUTCOME MEASURES:

1. Primary Outcome: Verbal Pain Score
Description: 11 point verbal pain score (VPS) 0=no pain; 10=worst imaginable pain
Time Frame: Immediately after injection of study drug. One time assessment.
Measure: Median (Inter-Quartile Range); unit: Units on a scale
Arm/Group | Control Arm | Lidocaine / Propofol Admixture Arm | Lidocaine Pretreatment Arm
Number analyzed (Participants) | 50 | 50 | 51
Units on a scale | 3 [0 to 6] | 0 [0 to 2] | 0 [0 to 0]
Statistical Analysis 1: Comparison: Control Arm vs Lidocaine / Propofol Admixture Arm vs Lidocaine Pretreatment Arm; Hypothesis: Lidocaine / propofol admixture would be superior to lidocaine pretreatment for attenuating propofol-induced injection pain. Sample size calculated to detect a difference of at least 2 VPS points; beta 0.8; Test type: Superiority or Other; p < 0.0001, Kruskal-Wallis

2. Secondary Outcome: Complete Alleviation of Injection Pain
Description: Total subjects within the arm versus those subjects who had no pain with injection (VPS=0)
Time Frame: Immediately after injection of study drug. One time assessment
Measure: Number; unit: Participants
Arm/Group | Control Arm | Lidocaine / Propofol Admixture Arm | Lidocaine Pretreatment Arm
Number analyzed (Participants) | 50 | 50 | 51
Participants | 14 | 28 | 40
Statistical Analysis 1: Comparison: Control Arm vs Lidocaine / Propofol Admixture Arm vs Lidocaine Pretreatment Arm; Test type: Superiority or Other; p < 0.008, Chi-squared; Fisher's exact test after chi-squared

3. Secondary Outcome: Satisfaction With Anesthetic Technique
Description: Were you satisfied with the anesthetic technique? Yes/No
Time Frame: Prior to discharge. One time assessment
Measure: Number; unit: Participants
Arm/Group | Control Arm | Lidocaine / Propofol Admixture Arm | Lidocaine Pretreatment Arm
Number analyzed (Participants) | 50 | 50 | 51
Participants
  Yes | 42 | 48 | 51
  No | 8 | 2 | 0

ADVERSE EVENTS:
Arm/Group | Control Arm | Lidocaine / Propofol Admixture Arm | Lidocaine Pretreatment Arm
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/51 | 0/53
Other Adverse Events (participants affected / at risk) | 0/52 | 0/51 | 0/53

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No